CLINICAL TRIAL: NCT06411158
Title: Training for Urinary Leakage Improvement After Pregnancy
Acronym: TULIP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NICHD Pelvic Floor Disorders Network (Network)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Duke University (Other); Kaiser Permanente (Other); University of California, San Diego (Other); University of Chicago (Other); University of Pennsylvania (Other); University of Texas Southwestern Medical Center (Other); Women and Infants Hospital of Rhode Island (Other); RTI International (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PFDN-32P01; UG1HD069013 (NIH); UG1HD054214 (NIH); UG1HD041267 (NIH); UG1HD054241 (NIH); UG1HD110057 (NIH); UG1HD069010 (NIH); U24HD069031 (NIH)
Record Dates: First submitted 2024-05-03; First posted 2024-05-13 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Urinary Incontinence; Delivery Complication
Keywords: Urinary Incontinence; Pelvic Floor Disorders; Physical Therapy; Biofeedback; Anal Incontinence
MeSH Terms: conditions — Urinary Incontinence; Pelvic Floor Disorders; Encopresis | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: The primary analyses will use an intention-to-treat (ITT) population to compare change from baseline in ICIQ-SF score at 6 months between treatment groups using a general linear mixed model.
Who Masked: Outcomes Assessor
Masking Description: The primary outcome will be assessed at 6 months postpartum by blinded outcomes assessors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Interventionist-guided training (Active Comparator): Interventionist-guided training at baseline (i.e., approximately 8 weeks postpartum), followed by a Home Exercise Prescription (HEP), a second interventionist-guided training session approximately 4 weeks later, and then continued HEP. Two exercise sets per day are encouraged between baseline and 6 months postpartum (i.e., time of the primary outcome), followed by at least 3 times-per-week exercise sets until 12 months postpartum. Home exercises will be encouraged using a PFDN research smartphone app, resources to help participants with home exercises and prompts for participants to confirm the number of exercise sets completed.
  Interventions: Other: Interventionist-guided training
- Home pelvic floor exercises guided by the leva® device (Active Comparator): Home pelvic floor exercises guided by the leva® device and its accompanying app/software for gradually increasing strength and duration of pelvic floor contractions. The PFDN research smartphone app will have weekly queries of whether exercises were completed.
  Interventions: Device: Home pelvic floor exercises guided by the leva® device
- Education (Other): Education will be provided on pelvic floor muscle function and continence mechanisms. No specific prescription or verbal direction will be given regarding the suggested number and frequency of home pelvic floor muscle exercises.
  Interventions: Other: Education

INTERVENTIONS:
Other: Interventionist-guided training — Interventionist-guided training at baseline (i.e., approximately 6 weeks postpartum), followed by a Home Exercise Prescription (HEP), a second interventionist-guided training session approximately 4 weeks later, and then continued HEP. Two exercise sets per day are encouraged between baseline and 6 months postpartum (i.e., time of the primary outcome), followed by at least 3 times-per-week exercise sets until 12 months postpartum. Home exercises will be encouraged using a PFDN research smartphone app, resources to help participants with home exercises and prompts for participants to confirm the number of exercise sets completed.
  Arms: Interventionist-guided training
Device: Home pelvic floor exercises guided by the leva® device — Home pelvic floor exercises guided by the leva® device and its accompanying app/software for gradually increasing strength and duration of pelvic floor contractions. Between baseline and 6 months postpartum, twice-daily exercise sets will be encouraged, followed by at least 3 times-per-week exercises from 6 to 12 months postpartum. As in Arm 1, the PFDN research smartphone app, resources to help participants with home exercises and prompts for participants to confirm the number of exercise sets completed.
  Arms: Home pelvic floor exercises guided by the leva® device
Other: Education — Education will be provided on pelvic floor muscle function and continence mechanisms. No specific prescription or verbal direction will be given regarding the suggested number and frequency of home pelvic floor muscle exercises.
  Arms: Education

SUMMARY:
This is a multi-center, randomized single-blind nonsurgical trial conducted in approximately 216 primiparous postpartum women at high risk for prolonged/sustained pelvic floor disorders with symptomatic, bothersome urinary incontinence (UI) amenable to nonsurgical treatment.

TULIP is a 3-Arm trial with two active interventions (Arms 1 and 2) and a Patient Education control arm (Arm 3). Arm 1 consists of pelvic floor muscle training (PFMT). Arm 2 uses a home biofeedback device (leva®).

The primary outcome will be assessed at 6 months postpartum by blinded outcomes assessors, and follow-up will continue until 12 months postpartum.

DETAILED DESCRIPTION:
TULIP is a 3-Arm trial with two active interventions (Arms 1 and 2) and a Patient Education control arm (Arm 3). Arm 1 consists of pelvic floor muscle training (PFMT) sessions with a skilled interventionist. Arm 2 uses a home biofeedback device (leva®).

All groups will have access to basic education on stress urinary incontinence, overactive bladder, pelvic floor muscle function and continence mechanisms.

Arm 1 will consist of interventionist-guided training at baseline (approximately 8 weeks postpartum), followed by a Home Exercise Prescription (HEP), a second interventionist-guided training session (approximately 4 weeks later), and then continued HEP until 12 months postpartum. Home exercises will be encouraged using a PFDN research smartphone app, resources to help participants with home exercises and prompts for participants to confirm the number of exercise sets completed.

Arm 2 will consist of home pelvic floor exercises guided by the leva® device and its accompanying app/software for gradually increasing strength and duration of pelvic floor contractions. The Arm 2 exercise regimen begins at approximately 8 weeks postpartum and continues until 12 months postpartum. As in Arm 1, the PFDN research smartphone app resources to help participants with home exercises and prompts for participants to confirm the number of exercise sets completed.

Arm 3 participants will only be provided basic education materials. No specific prescription or verbal direction will be given regarding the suggested number and frequency of home pelvic floor muscle exercises.

The primary outcome is change in UI as measured by the ICIQ-SF, comparing scores from baseline to 6 months postpartum. The questionnaire will be sent to participants monthly from baseline through 12 months postpartum, and change through 12 months postpartum is a secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18yo primiparous patient s/p singleton vaginal delivery (>32 weeks), approximately 6wk postpartum
2. At increased risk of sustained pelvic floor disorders, as defined by

   1. neonate ≥3.5kg, and/or
   2. operative delivery (i.e., forceps or vacuum-assisted vaginal delivery), and/or
   3. ≥2nd-degree perineal laceration
3. Symptomatic, bothersome UI as defined by a score of ≥6 on the ICIQ-SF.

Exclusion Criteria:

1. Inability to complete study assessments or procedures, per clinician judgment, or not available for 6mo postpartum follow-up
2. Stillbirth or significant maternal or neonatal illness
3. Non-English or non-Spanish speaking
4. Perineal wound breakdown or cloaca observed on exam
5. Severe pain with assessments of PFM integrity and/or strength/function
6. Already engaged (since delivery) in in-person physical therapy for strengthening of the pelvic floor
7. Unwilling or unable to upload and use external smartphone app(s)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 216 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2027-05-12 (Estimated); Study Completion 2027-11-12 (Estimated)

PRIMARY OUTCOMES:
Change in urinary incontinence measure by the ICIQ-SF | From baseline to 6 months postpartum
  The primary outcome is change in urinary incontinence (UI) as measured by the International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF), comparing scores from baseline to 6 months postpartum. This instrument consists of 3 scorable questions measuring frequency of leakage, volume of leakage, and associated bother with leakage. ICIQ-SF scores range from 0 (no leakage or bother) to 21 (worst leakage, most bothersome).

SECONDARY OUTCOMES:
Change in Lower Urinary Tract Dysfunction Research Network Symptom Index (LURN-SI-10) score | From baseline to 6 months and 12 months postpartum
  Lower Urinary Tract Dysfunction Research Network Symptom Index (LURN-SI-10) is designed to address a broader spectrum of lower urinary tract symptoms, particularly incontinence, bladder pain, and post-micturition symptoms. The LURN-SI-10 score ranges from 0 (least severe) to 38 (most severe).
Patient Global Impression of Improvement (PGI-I) score | At 6 months and 12 months postpartum
  Patient Global Impression of Improvement (PGI-I) captures a participant's perceived improvement from baseline, defined as (1) = very much better, (2) = much better, (3) = a little better, (4) = no change, (5) = a little worse, (6) much worse, (7) very much worse.
Change in St. Mark's score | From baseline to 6 months and 12 months postpartum
  The St. Mark's questionnaire is used to assess anal incontinence symptom severity. St. Mark's Score, ranges from 0 (perfect fecal continence) to 24 (total fecal incontinence).
Female Sexual Function Index (FSFI) score | At 6 months and 12 months postpartum
  Sexual function will be assessed using the Female Sexual Function Index (FSFI), which uses 19 questions to measure 6 domains: desire, arousal, lubrication, orgasm, satisfaction, and pain. Female Sexual Function Index scores range from 2.0 (lowest sexual function) to 36.0 (high sexual function).
Change in urinary incontinence measure by the ICIQ-SF | From baseline to 12 months postpartum
  The International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF) consists of 3 scorable questions measuring frequency of leakage, volume of leakage, and associated bother with leakage. ICIQ-SF scores range from 0 (no leakage or bother) to 21 (worst leakage, most bothersome).

CONTACTS AND LOCATIONS:
Overall Officials: David Rahn, MD, Principal Investigator — UTSW; Marie Gantz, PhD, Principal Investigator — RTI International
Locations (7):
- United States (7):
  - Kaiser Permanente -- San Diego, San Diego, California
  - University of California - San Diego, San Diego, California
  - University of Chicago, Chicago, Illinois
  - Duke University, Duke Division of Urogynecology and Reconstructive Pelvic Surgery, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Brown/ Women and Infants Hospital of Rhode Island, Center for Women's Pelvic Medicine and Reconstructive Surgery, Providence, Rhode Island
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Study data will be made available through DASH
Time Frame: Plan to submit full study dataset before the end of the award period.
Access Criteria: Access is managed by DASH.
URL: http://dash.nichd.nih.gov/